CLINICAL TRIAL: NCT04708314
Title: An Open-Label Study to Evaluate the Safety of Golodirsen in Non-Ambulant Patients With Duchenne Muscular Dystrophy
Brief Title: An Open-Label Study of Golodirsen in Non-Ambulant Patients With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The Sponsor has decided to focus their resources on other areas of therapy.
Sponsor: Rare Disease Research, LLC (Other)
Collaborators: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-06-001
Record Dates: First submitted 2020-09-21; First posted 2021-01-13 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — golodirsen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 30 mg/kg (Other): Golodirsen 30 mg/kg will be administered as an intravenous (IV) infusion over approximately 35 to 60 minutes once a week during the treatment period (up to 96 weeks). After the treatment period, patients can go into a safety extension period (not to exceed 48 weeks) until the patient is able to transition to commercially available drug or a separate golodirsen study.
  Interventions: Drug: Golodirsen 50 MG/1 ML Intravenous Solution [VYONDYS 53]

INTERVENTIONS:
Drug: Golodirsen 50 MG/1 ML Intravenous Solution [VYONDYS 53] — Vyondys 53

SUMMARY:
This is an open-label study to evaluate the safety and tolerability of golodirsen injection in Non-ambulant DMD patients with confirmed genetic mutations amenable to treatment by exon 53 skipping (Golodirsen).

Golodirsen 30 mg/kg will be administered as an intravenous (IV) infusion over approximately 35 to 60 minutes once a week during the treatment period (up to 96 weeks). After the treatment period, patients can go into a safety extension period (not to exceed 48 weeks) until the patient is able to transition to commercially available drug or a separate golodirsen study.

Safety will be regularly assessed throughout the study via the collection of adverse events (AEs), laboratory tests, electrocardiograms (ECGs), echocardiograms (ECHOs), vital signs, and physical examinations. Exploratory assessments, including pulmonary function tests (PFTs), upper extremity testing, and other measurements of functional status, will occur at functional assessment visits every 12 weeks over the first year of treatment and approximately every 24 weeks over the second year of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male with DMD with a mutation that may be amenable to exon 53 skipping as documented by a genetic report from an accredited laboratory confirming mutation endpoints by multiplex ligation-dependent probe amplification.
2. Be 7 years of age or older.
3. Has been on a stable dose of oral corticosteroids for at least 24 weeks prior to study drug administration and the dose is expected to remain constant (except for modifications to accommodate changes in weight) throughout the study or has not received corticosteroids for at least 24 weeks prior to study drug administration and does not expect to start corticosteroids throughout the study.
4. Be unable to ambulate ("non-ambulatory"). By definition, loss of ambulation means patient or caregiver reported continuous wheelchair use that has been verified by a clinical evaluator. The following conditions should be met:

   1. Condition is not secondary to acute worsening of mobility due to orthopedic morbidity (eg, fracture, sprain, or injury) or surgical procedure.
   2. Unable to perform 10-meter walk run test.
5. Has stable pulmonary function that, in the opinion of the Investigator, is unlikely to decompensate over the study period.
6. Patients who are post-pubertal and sexually active must agree to use, for the entire duration of the study and for 90 days post last dose, a male condom and the female sexual partner must also use a medically acceptable form of birth control (eg, oral contraceptives).
7. Able to understand and comply with all study requirements, in the Investigator's opinion, or if under the age of 18 years, must have a parent(s) or legal guardian(s) who is able to understand.
8. Willing to provide informed consent to participate in the study, or if under the age of 18 years, be willing to provide informed assent, if applicable, and have a parent(s) or legal guardian(s) who is willing to provide informed consent for the patient to participate in the study.

Exclusion Criteria:

1. Use of any pharmacologic treatment (other than corticosteroids) within 12 weeks of study drug administration that in the opinion of the Investigator might have an effect on skeletal muscle strength or function (eg, growth hormone, anabolic steroids).
2. Previous treatment with any investigational drug or exon skipping therapy within the last 3 months.
3. Major change in physiotherapy regimen within the past 3 months or expected change over the study period.
4. Major surgery within 3 months of study drug administration or planned major surgery for any time during this study.
5. Presence of other clinically significant illness that cannot be attributed to classic Duchenne disease course including significant cardiac, pulmonary, hepatic, renal, hematologic, immunologic, behavioral disease, or malignancy.
6. Systemic use of any aminoglycoside antibiotic within 12 weeks of study drug administration or anticipated need for use of an aminoglycoside antibiotic or statin during the study.
7. Must not require antiarrhythmic and/or antidiuretic therapy for heart failure. Patients are allowed to take other medication including angiotensin-converting enzyme (ACE) inhibitors, angiotensin receptor blocking agents, β blockers or potassium, provided they have been on a stable dose for 24 weeks prior to study drug administration and the dose is expected to remain constant throughout the study.
8. If the patient is asymptomatic but has a LVEF < 40% at Screening or clinically significant at the discretion of Investigator, the Investigator should discuss inclusion of patient in the study with the appropriate institutional safety committee or medical monitor.
9. Prior or ongoing medical condition that could, in the Investigator's opinion, adversely affect the safety of the patient, make it unlikely that the course of treatment would be completed, or impair the assessment of study results.

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only male patients are affected by this condition
Enrollment: 2 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Explore the safety and tolerability of Golodirsen in number of participants with Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs | Baseline up to 96 weeks
  Adverse Event (AE) was any untoward medical occurrence in a participant that did not necessarily have a causal relationship with the study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death; Life-threatening event; required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Treatment emergent adverse events were events that developed or worsened during the on-treatment period (defined as time from first dose of study drug and up to 28 days after last dose of study drug [up to 148 weeks]) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.

OTHER OUTCOMES:
Change from Baseline to Week 96 in Forced Vital Capacity Percent (FVC%) Predicted | Baseline up to 96 weeks
  FVC is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry; and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes. Percent of predicted FVC = (observed value) / (predicted value) * 100%.
Change from Baseline to Week 96 in Performance of Upper Limb (PUL) Score | Baseline up to 96 weeks
  The PUL was specifically designed for DMD patients to evaluate the progression of weakness and natural history of functional decline in DMD. Psychometric methods were employed to create a viable scale to enable a clinician-reported outcome assessment tool that can establish clinical meaningfulness and relevance of activities of daily living (ADL).
Change from Baseline to Week 96 in Brooke scale for upper extremity | Baseline up to 96 weeks
  The Brooke Score for Arms and Shoulders was developed specifically for use in this population to assess arm and shoulder function over 6 functional grades.
Change from Baseline to Week 96 in 9-Hole Peg Test | Baseline up to 96 weeks
  In this timed test, the patient is instructed to take 9 pegs from a shallow bowl in the testing apparatus and put each peg into a hole, 1 at a time. When all 9 pegs are in place, the patient takes them out 1 at a time and puts them back in the shallow bowl. This test is repeated twice with each hand and the best time for each hand is recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania